CLINICAL TRIAL: NCT00303706
Title: A Prospective Randomized Trial of Endoscopic Versus Conventional Harvesting of the Radial Artery in Coronary Artery Bypass
Brief Title: Study of Endoscopic Versus Open Harvest of the Radial Artery in Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Johnson & Johnson (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-05-053
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
Keywords: CABG, Endoscopic, Radial Artery; Radial Artery Conduit; Coronary Artery Bypass Surgery; Endoscopic technique
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: Endoscopic Radial Artery Harvest

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of minimally invasive endoscopic harvest of the radial artery to the conventional open method of radial artery harvest in coronary artery bypass surgery. The researchers hypothesize that the radial artery can be safely, efficiently, and routinely harvested using a minimally invasive endoscopic technique. Endoscopic minimally invasive harvesting of the radial artery will reduce the postoperative morbidity due to pain, wound infection, and neurological complications and improve cosmetic results.

DETAILED DESCRIPTION:
Many surgical disciplines have been quick to adopt minimally invasive techniques because of decreased complications and shorter recovery times. As we enter the fifth decade of coronary artery bypass grafting surgery more attempts are being made to perform the operation less invasively. Harvesting of the saphenous vein (a large superficial vein in the leg which is routinely used in bypass surgery) using a telescope (camera), has been shown to be superior to harvesting the vein through a large open incision. At our institution, this vein mentioned above, is routinely harvested using less invasive techniques with a camera. This has been shown to result in less infection.

In the early 1990's, the radial artery was reintroduced into bypass surgery to increase the number of available alternative bypass grafts. Long-term results of the radial artery (8-9 years) have shown that 88-91% of the radial arteries harvested remain open thereby allowing the flow of blood. This is significantly better than the 10-year rates of the saphenous vein of 53-67%. Therefore, the radial artery has become more popular as a bypass graft.

Conventionally, the radial artery is harvested by making a long vertical incision extending from the wrist to the elbow. The radial artery is then dissected under direct vision within this large open incision. Complications from the open harvest of the radial artery include infection, neurological complications, possible decrease blood flow to the hand, and poor wound healing or scarring.

Recently, with the development of endoscopic harvesting systems, the radial artery can be harvested using a telescope (camera) and very small incisions. Thus far, to our knowledge there have been no published studies comparing conventional techniques to less invasive endoscopic techniques for harvesting the radial artery. Therefore, we propose a prospective randomized study to determine if the radial artery can be routinely harvested using an endoscopic minimally invasive technique. We wish to compare the conventional open technique to the minimally invasive technique to determine if there are any differences in postoperative complications, length of hospital stay or possible differences in patient satisfaction in cosmetic results (scarring) between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients greater than 18 years of age with coronary artery disease requiring elective, urgent, or emergency coronary artery revascularization where the radial artery can be used as a bypass conduit.

Exclusion Criteria:

* Patient's refusal to have surgery, inability to give informed consent, and contraindication in harvesting the radial artery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2005-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome event will be the rate of forearm wound infection at 6 weeks. | 6 weeks

SECONDARY OUTCOMES:
Wound pain | 6 weeks
Neurological complications | 6 weeks
Patient satisfaction | 6 weeks
Length of hospitalization | will vary with patient lenght of stay
Histological integrity of the harvested radial artery | during OR

CONTACTS AND LOCATIONS:
Overall Officials: Bob Kiaii, MD, FRCSC, Principal Investigator — Department of Cardiac Surgery, University of Western Ontario and the London Health Sciences Centre, University Hospital
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Kiaii B, Moon BC, Massel D, Langlois Y, Austin TW, Willoughby A, Guiraudon C, Howard CR, Guo LR. A prospective randomized trial of endoscopic versus conventional harvesting of the saphenous vein in coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2002 Feb;123(2):204-12. doi: 10.1067/mtc.2002.118682. PMID 11828277
- [Background] Possati G, Gaudino M, Prati F, Alessandrini F, Trani C, Glieca F, Mazzari MA, Luciani N, Schiavoni G. Long-term results of the radial artery used for myocardial revascularization. Circulation. 2003 Sep 16;108(11):1350-4. doi: 10.1161/01.CIR.0000087402.13786.D0. Epub 2003 Aug 25. PMID 12939220
- [Background] Trick WE, Scheckler WE, Tokars JI, Jones KC, Smith EM, Reppen ML, Jarvis WR. Risk factors for radial artery harvest site infection following coronary artery bypass graft surgery. Clin Infect Dis. 2000 Feb;30(2):270-5. doi: 10.1086/313657. PMID 10671327
- [Background] Brodman RF, Frame R, Camacho M, Hu E, Chen A, Hollinger I. Routine use of unilateral and bilateral radial arteries for coronary artery bypass graft surgery. J Am Coll Cardiol. 1996 Oct;28(4):959-63. doi: 10.1016/s0735-1097(96)00265-3. PMID 8837574
- [Background] Denton TA, Trento L, Cohen M, Kass RM, Blanche C, Raissi S, Cheng W, Fontana GP, Trento A. Radial artery harvesting for coronary bypass operations: neurologic complications and their potential mechanisms. J Thorac Cardiovasc Surg. 2001 May;121(5):951-6. doi: 10.1067/mtc.2001.112833. PMID 11326239
- [Background] Dumanian GA, Segalman K, Mispireta LA, Walsh JA, Hendrickson MF, Wilgis EF. Radial artery use in bypass grafting does not change digital blood flow or hand function. Ann Thorac Surg. 1998 May;65(5):1284-7. doi: 10.1016/s0003-4975(98)00176-3. PMID 9594852
- [Background] Serricchio M, Gaudino M, Tondi P, Gasbarrini A, Gerardino L, Santoliquido A, Pola P, Possati G. Hemodynamic and functional consequences of radial artery removal for coronary artery bypass grafting. Am J Cardiol. 1999 Dec 1;84(11):1353-6, A8. doi: 10.1016/s0002-9149(99)00573-1. PMID 10614806
- [Background] Connolly MW, Torrillo LD, Stauder MJ, Patel NU, McCabe JC, Loulmet DF, Subramanian VA. Endoscopic radial artery harvesting: results of first 300 patients. Ann Thorac Surg. 2002 Aug;74(2):502-5; discussion 506. doi: 10.1016/s0003-4975(02)03717-7. PMID 12173836